CLINICAL TRIAL: NCT06830902
Title: Comparison of Stent Related Symptoms Between Regular Double J Stent Versus Comfi J Stent: A Single Blinded Randomized Controlled Trial
Brief Title: Comparison of Stent-Related Symptoms: Regular Double J Stent vs. Comfi J Stent
Acronym: COMFIJ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bir Hospital (Other Government)
Collaborators: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Anil Shrestha, Professor Dr., Bir Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ComfiJ
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Stent Related Symptoms

STUDY DESIGN:
Intervention Model Description: Single Blind, Randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regular Double J stent (Active Comparator): Regular Double J stent placement
  Interventions: Device: Regular Double J stent
- Comfi J stent (Active Comparator): Comfi J stent placement
  Interventions: Device: Comfi J stent

INTERVENTIONS:
Device: Regular Double J stent — Regular Double J stent
  Arms: Regular Double J stent
Device: Comfi J stent — Comfi J stent
  Arms: Comfi J stent

SUMMARY:
A prospective, single-blinded, randomized controlled trial conducted at a single center to compare stent related symptoms between two different stents using Ureteral Stent Symptom Questionnaire (USSQ) scores , Visual Analog Scale (VAS) pain scores.

DETAILED DESCRIPTION:
Ureteral stents are widely used in urology following retrograde intrarenal surgeries and ureteric lithotripsy and other endourological procedures. However, their use is associated with significant discomfort, infections, and reduced quality of life (QoL). Over time, different materials and designs have been developed to improve stent performance and reduce complications. This study aims to compare the stent-related symptoms (SRS) of two types of ureteral stents: the regular Double J stent and the Comfi J stent.

Objectives of the study-

1. Compare Ureteral Stent Symptom Questionnaire (USSQ) scores between the two stents.
2. Compare Visual Analog Scale (VAS) pain scores.
3. Assess complications associated with each stent.
4. Evaluate the difficulty of stent insertion.

Study Design & Methods: A prospective, single-blinded, randomized controlled trial conducted at a single center. Sample Size: 100 patients undergoing retrograde intrarenal surgery, ureteroscopic lithotripsy

Randomization: Intraoperative, using a computer-generated sequence, block randomization Assessments: USSQ and VAS scores at post-operative days (POD) 1, 7, and 14.

Statistical Analysis: Statistical Package for the Social Sciences software with a significance threshold of p < 0.05.

Expected Outcomes: Determining whether the Comfi J stent reduces pain, urinary symptoms, and other complications compared to the regular Double J stent.

Evaluating if changes in design/material can improve patient QoL.

Ethical Considerations:

Institutional ethics approval and informed consent from all participants. Confidentiality ensured, with voluntary participation.

This study aims to provide evidence-based recommendations for improving ureteral stent tolerability and reducing patient morbidity

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were adult patients (aged 18-80 years) who underwent unilateral retrograde ureteroscopy (URS) lithotripsy for stone disease
* Retrograde intrarenal surgery (RIRS) lithotripsy with planned ureteric stent insertion for urinary tract stones

Exclusion Criteria:

* Concomitant use of a-blockers, anticholinergics, corticosteroids, calcium channel blockers, and analgesics
* Undergoing percutaneous nephrolithotomy, open ureteric surgery or laparoscopic ureteric surgery, including ureterolithotomy
* Neurogenic bladder, Overactive bladder syndrome, and neurological and psychiatric diseases
* Preoperative febrile Urinary Tract Infection (UTI)
* Pregnancy or breastfeeding;
* A single kidney
* Moderate or severe cardiovascular or cerebrovascular disease
* Hepatic dysfunction
* History of pelvic surgery or irradiation
* History of bladder or prostate surgery
* Other acute medical conditions (including acute pancreatitis, acute gastroenteritis, musculoskeletal disorders) that might influence the USSQ pain score
* Allergy to any medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Stent related symptom | 2 weeks
  Comparison of Ureteral Stent Symptom Questionnaire (USSQ) scores between regular Double J stent and Comfi J stent at postoperative day 1, 7, and 14. Higher Scores means greater severity of the symptoms.

SECONDARY OUTCOMES:
Complication rates | before 2 weeks
  Incidence of stent-related complications such as fever, stent migration, expulsion, or readmission. Early removal of stent due to stent related symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Bir Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No